CLINICAL TRIAL: NCT05519111
Title: Dronabinol for the Reduction of Chronic Pain and Inflammation in People With Sickle Cell Disease
Brief Title: Cannabinoids for the Reduction of Inflammation and Sickle Cell Related Pain
Acronym: CRISP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Susanna Curtis, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GCO 22-1141; K23HL151884 (NIH)
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to dronabinol or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Dronabinol and placebo will be over-encapsulated so that neither participants nor investigators are aware of the subjects assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dronabinol (Experimental): BID for 8 weeks. Dosage will be individualized per patient. In days 1-4 of the study each patient will be titrated from 5mg bid to a minimum dose of 2.5 mg bid to a maximum dose of 10 mg bid depending on patient preference.
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator): A placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Dronabinol, an FDA approval oral agent containing synthetic tetrahydrocannabinol (THC)
  Other Names: Marinol
  Arms: Dronabinol
Drug: Placebo — placebo equivalent
  Arms: Placebo

SUMMARY:
A randomized, double blind, study of dronabinol as a palliative agent in the treatment of pain, inflammation, and other complications of sickle cell disease (SCD).

DETAILED DESCRIPTION:
A randomized, double blind, study of dronabinol as a palliative agent in the treatment of pain, inflammation, and other complications of sickle cell disease (SCD).

Primary Objective: To determine whether dronabinol will improve pain and QOL in adults with SCD and chronic pain.

Secondary Objectives: To assess dronabinol's effect on markers of inflammation in patients with SCD compared to placebo.

To determine the safety and tolerability of dronabinol use in adults with SCD compared to placebo.

ELIGIBILITY:
* Age >18 years
* Clinical diagnosis of SCD (HbSS, HbSC, HbSβ+; Thal, HbSβ0Thal, HbS variants)
* Baseline score of 60 or lower on the ASCQ-Me 7-day pain interference domain
* If on a SCD modifying therapy (hydroxyurea, regular blood transfusions, L-glutamine, voxelotor, crizanlizumab), on stable dose for at least 3 months
* If using opioids for pain at home, on stable dose for at least 3 months
* One urine toxicology negative for cannabinoids within 30 days of randomization
* No known intolerance to dronabinol, or marijuana
* No history of psychotic episode, psychosis, or active suicidality
* No contraindication to dronabinol with attention to potential side effects, concurrent medications/substances, and concurrent medical problems, as evaluated by a physician
* Willing to abstain from cannabis, medical and illicit, during study weeks 1 through 8
* Not pregnant or nursing
* If a woman capable of becoming pregnant, willing to use a medically accepted form of birth control for the duration of study participation. Accepted forms include oral contraception, medroxyprogesterone, contraceptive implants or patch, surgical sterilization, total abstinence.
* Able to consent for research
* No daily cannabis use
* No diagnosis of active substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Measurement Outcome Information System (PROMIS) pain impact score | end of study at 8 weeks
  Change in Patient Reported Measurement Outcome Information System (PROMIS) pain impact score. Total scale from 20-80, median of 50 and SD of 10. Higher score represent poorer health outcomes.

SECONDARY OUTCOMES:
Adult Sickle Cell Quality of Life Information System (ASCQ-Me) Pain impact | end of study at 8 weeks
  Total scale from 20 to 80, median of 50 and SD of 10. Higher scores represent better health outcomes.
Quality of Life Outcomes | end of study at 8 weeks
  ASCQ-Me survey domains for emotional impact, social impact, stiffness, and sleep.
  Each domain scale from 20 to 80, median of 50 and SD of 10. Higher scores represent better health outcomes.
  Total scale from 20 to 80, median of 50 and SD of 10. Higher scores represent better health outcomes.
WBC with differential | end of study at 8 weeks
  a marker of Inflammation. The blood differential test measures the percentage of each type of white blood cell (WBC) in the blood. It also reveals if there are any abnormal or immature cells.
C-reactive protein (CRP) | end of study at 8 weeks
  marker of Inflammation. C-reactive protein (CRP) is produced by the liver. The level of CRP rises when there is inflammation throughout the body. It is one of a group of proteins, called acute phase reactants, that go up in response to inflammation. The levels of acute phase reactants increase in response to certain inflammatory proteins called cytokines. These proteins are produced by white blood cells during inflammation.
tryptase | end of study at 8 weeks
  marker of Inflammation. tryptase is an enzyme found in mast cells
substance P | end of study at 8 weeks
  marker of Inflammation. Substance P ("P" standing for "Preparation" or "Powder") is a neuropeptide - but only nominally so, as it is ubiquitous. Its receptor - the neurokinin type 1 - is distributed over cytoplasmic membranes of many cell types (neurons, glia, endothelia of capillaries and lymphatics, fibroblasts, stem cells, white blood cells) in many tissues and organs. SP amplifies or excites most cellular processes.
Vascular cell adhesion protein 1 (VCAM-1) | end of study at 8 weeks
  marker of Inflammation. plasma levels of oxidative stress and adhesion molecules
cytokine IL1a | end of study at 8 weeks
  marker of Inflammation. Interleukin 1 alpha (IL-1α) also known as hematopoietin 1 is a cytokine of the interleukin 1 family that in humans is encoded by the IL1A gene.
cytokine IL1b | end of study at 8 weeks
  marker of Inflammation. Interleukin 1 beta (IL-1β) also known as leukocytic pyrogen, leukocytic endogenous mediator, mononuclear cell factor, lymphocyte activating factor and other names, is a cytokine protein that in humans is encoded by the IL1B gene.
cytokine IL6 | end of study at 8 weeks
  marker of Inflammation. Interleukin-6 (IL-6) is a pleiotropic cytokine with central roles in immune regulation, inflammation, hematopoiesis, and oncogenesis.
cytokine IL4 | end of study at 8 weeks
  marker of Inflammation. The interleukin 4 (IL4, IL-4) is a cytokine that induces differentiation of naive helper T cells (Th0 cells) to Th2 cells.
cytokine IL10 | end of study at 8 weeks
  marker of Inflammation. Interleukin 10 (IL-10), also known as human cytokine synthesis inhibitory factor (CSIF), is an anti-inflammatory cytokine.
tumor necrosis factor alpha (TNFα). | end of study at 8 weeks
  marker of Inflammation. Tumor necrosis factor (TNF), a 17 kDa protein consisting of 157 amino acids, is a homotrimer in solution that is mainly produced by activated macrophages, T lymphocytes, and natural killer (NK) cells.
PROMIS domains | end of study at 8 weeks
  PROMIS domains for anxiety, appetite, nausea, and cognitive function, opioid use in oral morphine equivalents (OME), episodes of emergency room, hospital, or psychiatric facility utilization.
  Each domain scale from 20 to 80, median of 50 and SD of 10. Higher scores represent better health outcomes.
  Total scale from 20 to 80, median of 50 and SD of 10. Higher scores represent better health outcomes.
Columbia suicide severity rating scale | end of study at 8 weeks
  Columbia suicide severity rating scale. Full range from 0 to 9. Higher score represents higher intensity suicidal ideation.
Prodromal questionnaire brief version (PQ-B) | end of study at 8 weeks
  Prodromal questionnaire brief version: 21-item self-report instrument. Full scale range from 0 to 21, higher score represents poorer health outcomes
PROMIS domain for neuropathic pain quality | end of study at 8 weeks
  Total scale from 20-80, median of 50 and SD of 10. Higher scores represent worse outcomes.
PROMIS domain for nociceptive pain quality | end of study at 8 weeks
  Total scale from 20-80, median of 50 and SD of 10. Higher scores represent worse outcomes.
The Leeds assessment of neuropathic symptoms and signs (LANSS) Pain Scale | end of study at 8 weeks
  The Leeds assessment of neuropathic symptoms and signs (LANSS) Pain Scale comprises of a 7-item pain scale, including the sensory descriptors and items for sensory examination.
  Out of the seven items in the Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale (LANSS), five are symptom related and two are examination items.
  Full scale from scores between 0 and 24, higher score represents poorer health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Curtis, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Specify Other Time FrameOn request.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  Any purpose. Proposals should be directed to susanna.curtis@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (website tbd.)